CLINICAL TRIAL: NCT00397514
Title: Assessing the Hemodynamic Benefits of Cardiac Resynchronization Therapy in Children Following Open-Heart Surgery
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Shubhayan Sanatani, principal investigator, University of British Columbia
Other Study IDs: H03-70642; H03-70642 (Other: UBC)
Record Dates: First submitted 2006-11-07; First posted 2006-11-09 (Estimated); Results first posted 2013-08-30 (Estimated); Last update posted 2017-12-18 (Actual); Status verified 2017-11

CONDITIONS: Congenital Heart Defects
Keywords: Biventricular pacing; Congenital heart disease; Tissue Doppler echocardiography
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Congenital Heart Surgery Patients: Pacing protocol prior to patient's extubation with 20 min. of either conventional right ventricular (RV) or biventricular (BiV) pacing, preceded and followed by 10 min. of recovery time.
  Interventions: Procedure: Congenital Heart Surgery Patients

INTERVENTIONS:
Procedure: Congenital Heart Surgery Patients — undergoing either Biventricular (BiV) pacing or Right Ventricular (RV) Pacing

SUMMARY:
Malformations of the heart (congenital heart disease) are the most common congenital birth defects, occurring in about 1% of children. Each year, between 150-200 children will undergo open heart surgery at British Columbia Children's Hospital (BCCH) to repair the defect(s) in their heart. The abnormal structure of the heart or the open heart surgery may cause damage to the electrical system of the heart which can disturb the rhythm of the heart (arrhythmias), prolong recovery or be life-threatening. For this reason, temporary pacing wires are placed in the heart following surgery to ensure the heart rhythm is as normal as possible during the post-operative period (pacing). In recent years, scientists have recognized that pacing the heart from one area is not necessarily the same as pacing it from a different area. In fact, in some individuals with arrhythmias and poor heart function, pacing the heart from different areas can improve the pumping of the heart, resulting in better heart function. This form of treatment is called Cardiac Resynchronization Therapy (CRT) because it endeavours to optimize the pumping of the heart by changing the electrical activation of the heart. CRT has been used to a very limited extent in children. A few pediatric cardiologists have used CRT to help children who are in heart failure. We would like to determine whether pacing the heart from different areas after open heart surgery improves the child's heart function and aids his or her recovery.

DETAILED DESCRIPTION:
The heart's rhythmic beating or contraction is determined by the flow of an excitatory electrical wave-front along a specialized cardiac conduction system. In the presence of altered conduction, such as a bundle branch block or an intra-ventricular conduction delay, abnormal cardiac contraction or dyssynchrony occurs. The delay can occur in the specialized conduction system (electrical dyssynchrony) or myocardium (mechanical or structural dyssynchrony).1 Techniques to improve both electrical and mechanical synchrony in patients with bundle branch block were initially done on adults. Research in this field began to appear in the last decade when dual chamber pacing was first used as adjunctive therapy for adults with medically refractory heart failure.2 Acute studies showed that atrioventricular (AV) synchronous pacing with a short AV delay improved cardiac output and exercise duration in patients with heart failure and a prolonged PR interval.3 The beneficial effects of AV resynchrony (optimizing AV conduction times with pacing) were shown to be due to increased diastolic filling time, and reduction in mitral or tricuspid valve regurgitation. The results of long-term studies, however, did not demonstrate consistent improvement in ejection fraction or NYHA functional class with DDD pacing.4 Since then, Cardiac Resynchronization Therapy (CRT) has established itself as a proven therapy for congestive heart failure in adults, with patients showing improvement in exercise tolerance, quality of life, and survival.1, 5, 6 More recently, the technique of utilizing CRT to stimulate the heart from novel or multiple sites has been applied to pediatric patients.7-9 Children with chronic heart failure have received CRT successfully as an adjunctive therapy.

One of the major limitations of CRT is the objective assessment of whether cardiac output and ventricular function are improved. As well, the precise location of where to pace the heart in order to optimize hemodynamic function needs to be determined. The objective assessment of successful CRT is a difficult clinical issue and should ideally be performed non-invasively. Traditional two-dimensional echocardiographic and Doppler indices have been used to assess the efficacy of CRT and include measuring cardiac output, looking at ventricular ejection times, visually assessing wall motion, and measuring the length of diastole using the mitral "E" and "A" waves. As most of the existing techniques are limited to assessing global function, more detailed methods of assessment are necessary in order to fully assess and optimize CRT.10, 11 Tissue Doppler Imaging (TDI) offers a more detailed analysis of regional cardiac function and allows quantitative measures to be obtained. TDI operates at high frame rates and can non-invasively map cardiac activation and add information related to the degree and location of cardiac dyssychrony. TDI and its derivatives allow: (1) measurement of myocardial velocities, which is based on the detection of the Doppler shift caused by the motion of myocardial tissue during the cardiac cycle; (2) visualization of tissue tracking, which color-codes tissue segments with similar displacements according to a color map; (3) measurement of regional strain rates, which describes the rate of deformation, or how quickly a segment of tissue shortens or lengthens; and (4) measurement of regional strain, which describes the deformation of an object (in this case, tissue) relative to its original state. 12, 13

Cardiac pacing in children is done most often following cardiac surgery for congenital heart disease (CHD). This pacing is usually temporary. Following open heart surgery children frequently exhibit cardiac dyssynchrony secondary to conduction abnormalities or regional wall motion abnormalities. Often, damage to the conduction system is an unavoidable result of the operation itself. Regardless of the extent of the conduction abnormality, most patients operated on for congenital heart disease undergo a period of decreased cardiac function related to several factors, including: pre-existing myocardial disease; cardiopulmonary bypass; and residual cardiac lesions.7, 14 The decrease in cardiac performance and, therefore, the risk to the patient's life, can be aggravated by the presence of cardiac dyssynchrony. The benefits of CRT are just beginning to receive attention in the setting of pediatric post-operative cardiac care. 15

We hope to demonstrate that CRT is beneficial in the care of post-operative patients undergoing open-heart surgery for repair of congenital heart defects. We will be using state-of-the-art TDI for assessing cardiac dyssynchrony, and using it as a tool for monitoring therapy. This study has tremendous potential for application to all patients undergoing open-heart surgery for repair of congenital heart defects. If it can be demonstrated that CRT can improve post-operative outcomes in this population, significant morbidity and mortality can be avoided, Intensive Care Unit (ICU) and hospital stays shortened, and the associated health care costs reduced.

ELIGIBILITY:
Inclusion Criteria:

Subjects will be eligible for enrollment in this study if they are undergoing cardiopulmonary bypass surgery for right or left ventricular surgery or biventricular surgery and (1) have intra-cardiac conduction delay or bundle branch block post-surgery; (2) have echocardiographic evidence of ventricular dyssynchrony; (3) have pre-existing conduction disease or bundle branch block; or (4) have pre-existing ventricular dyssynchrony.

Exclusion Criteria:

Subjects will be excluded if they: (1) have single ventricle morphology; (2) require post-operative ECMO; (3) have sustained atrial or ventricular arrhythmias that may complicate ventricular pacing; (4) are not able to have functioning epicardial pacemaker leads; (5) are, in the opinion of the intensivist, cardiologist or surgeon, not stable enough medically to participate in the study; or (6) are unwilling to provide informed consent or assent.

Ages: 1 Week to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study cohort will consist of infants, children, and adolescents (<18 years) who are scheduled to undergo open-heart surgery for CHD. Each year approximately 150-200 patients undergo surgery to repair their CHD (see Section 6.4 for sample size estimates).
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2006-10; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shubhayan Sanatani, MD, Principal Investigator — Provincial Health Services Authority British Columbia
Locations (1):
- Children's Heart Centre, British Columbia's Children's Hospital, Vancouver, British Columbia, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 34 patients were recruited between October 1, 2006 and May 31, 2008.
Pre-assignment Details: One patient was excluded due to pacing wire malfunction. Four consented but we were not able to adequately capture and pace their left ventricle intraoperatively. Two consented, but underwent early extubation, and we were not able to perform the study in time. One family withdrew from the study. One patient had poor echocardiographic windows.
Groups:
- Congenital Heart Disease Pts. Undergoing Biventricular Repair: Pacing protocol prior to patient's extubation with 20 min. of conventional right ventricular (RV), preceded and followed by 10 min. of recovery time.
Period: Overall Study
Arm/Group | Congenital Heart Disease Pts. Undergoing Biventricular Repair
Started | 34
Completed | 25
Not Completed | 9
Not completed — Withdrawal by Subject | 1
Not completed — Pacing wire malfunction | 1
Not completed — Not able to capture & pace LV intraoper. | 4
Not completed — early extubation | 2
Not completed — poor echocardiographic windows | 1

BASELINE CHARACTERISTICS:
Population: The number of participants analyzed was 25 due to the withdrawal of 9 participants after enrolment as specified.
Groups:
- Congenital Heart Disease Patients: Pacing protocol prior to patient's extubation with 20 min. of conventional right ventricular (RV), preceded and followed by 10 min. of recovery time.
Arm/Group | Congenital Heart Disease Patients
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 25
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: months]
  Age, Continuous | 5.2 [0.1 to 37.4]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 11
Region of Enrollment [Number; unit: participants]
  Canada | 25

OUTCOME MEASURES:

1. Primary Outcome: Cardiac Index
Time Frame: Baseline and after 20 minutes of pacing
Measure: Median (Full Range); unit: L/min/m2
Groups:
- Baseline: Cardiac Index at baseline.
- BiV Pacing: Cardiac Index when patient's extubation with 20 min. of biventricular pacing
- RV Pacing: Cardiac Index when patient's extubation with 20 min. of right ventricular pacing
Arm/Group | Baseline | BiV Pacing | RV Pacing
Number analyzed (Participants) | 25 | 25 | 25
L/min/m2 | 3.39 [1.28 to 9.56] | 3.42 [1.03 to 8.40] | 3.23 [1.14 to 7.36]

2. Secondary Outcome: Systolic Blood Pressure
Reporting Status: Not Posted

3. Secondary Outcome: Incidence of Low Output Syndrome
Reporting Status: Not Posted

4. Secondary Outcome: TDI Indices (Tissue Velocities, Tissue Tracking, Regional Strain, and Regional Strain Rates)
Reporting Status: Not Posted

5. Secondary Outcome: Inotropic Support
Reporting Status: Not Posted

6. Secondary Outcome: Ventilatory Support
Reporting Status: Not Posted

7. Secondary Outcome: QRS Duration
Time Frame: Baseline and after 20 minutes of pacing
Measure: Median (Full Range); unit: ms
Groups:
- Baseline: QRS duration at baseline
- BiV Pacing: QRS duration when patient's extubation with 20 min. of biventricular pacing
- RV Pacing: QRS duration when patient's extubation with 20 min. of right ventricular pacing
Arm/Group | Baseline | BiV Pacing | RV Pacing
Number analyzed (Participants) | 25 | 25 | 25
ms | 80 [60 to 140] | 100 [80 to 100] | 100 [60 to 160]

8. Secondary Outcome: Cardio-pulmonary Bypass Time
Time Frame: Baseline and after 20 minutes
Measure: Median (Full Range); unit: min.
Arm/Group | Congenital Heart Disease Pts. Undergoing Biventricular Repair
Number analyzed (Participants) | 25
min. | 96 [55 to 236]

ADVERSE EVENTS:
Groups:
- Pacing Protocol and RV Pacing: Pacing protocol prior to patient's extubation with 20 min. of conventional right ventricular (RV), preceded and followed by 10 min. of recovery time.
Arm/Group | Pacing Protocol and RV Pacing
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 0/11

LIMITATIONS AND CAVEATS:
The study was limited by a small sample.Our study patients underwent BiV pacing just prior to extubation, by which time myocardial dysfunction may have recovered, so they represented a potentially healthier subset in comparison to adults.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No